CLINICAL TRIAL: NCT05115669
Title: Prospective, Open Clinical Investigation to Evaluate the Effectiveness and Safety of Wortie® Freeze Plus in the Treatment of Common Warts and Plantar Warts
Brief Title: Safety & Effectiveness of Wortie Freeze Plus in Common and Plantar Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karo Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E1573/WFP_001
Record Dates: First submitted 2021-10-15; First posted 2021-11-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Common Wart; Plantar Wart
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wortie freeze plus (Experimental): Cryogenic medical device (dimethylether-based product) + conductive gel + protective foam plasters.
  Up to 3 applications one every 14 days
  Interventions: Device: Wortie freeze plus

INTERVENTIONS:
Device: Wortie freeze plus — treatment of common and plantar warts

SUMMARY:
This is a Post-Market clinical Follow-up investigation to evaluate the safety and performed of the medical device Wortie Freeze Plus in the treatment of common and plantar warts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects.
2. Sex: male or female.
3. Age: 12 years old and above.
4. Subjects presenting at least 1 common wart (present since less than 6 months) on the fingers or back of the hands, and/or plantar wart (40-60% subjects with common wart) of a size less than 1 cm.
5. Subject, including minors having more than 12 years old, having given freely and expressly his/her informed consent.
6. Minor whose legally designated representative have given their free and express informed consent.
7. Subject affiliated to a health social security system.
8. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit, during all the study and at least 1 month after the study end

Exclusion Criteria:

1. Pregnant or nursing woman or planning a pregnancy during the study.
2. Subject who had been deprived of their freedom by administrative or legal decision.
3. Major subject who is under guardianship or who is not able to express his consent.
4. Subject in a social or sanitary establishment.
5. Subject suspected to be non-compliant according to the Investigator's judgment
6. Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
7. Subject with a cutaneous disease other than common warts, on the studied zone.
8. Subject with a known allergy to one of the components of the investigational device or conductive gel.
9. Subject who has diabetes.
10. Subject having problems with blood circulation or having a blood clotting condition.
11. Subject with immune deficiency or autoimmune disease.
12. Subject presenting more than 10 warts on the body
13. Subject presenting bleeding warts.
14. Subject presenting birthmarks, moles, warts with hairs growing from them, or any other spots on the treated and surrounding area.
15. Subject having a sensitive, inflamed, infected, irritated, red, damaged, cut, grazed, diseased or itchy skin on or around the treated zone.
16. Subject presenting genital warts, flat warts, filiform warts, periungual warts or warts with hairs growing from them.
17. Subject presenting 2 or more warts adjacent to each other
18. Subject undergoing a topical treatment on the test area or a systemic treatment: anti-inflammatory medication and/or antihistamines during the 2 weeks prior to screening and during the study; or corticosteroids during the 2 weeks prior to screening and during the study; or retinoids and/or immunosuppressors during the 3 months prior to screening and during the study; or any medication stabilized for less than a month
19. Subject who received a treatment of any type on the selected wart during the previous 6 months.
20. Subject having started or changed her oral contraceptive or any other hormonal treatment during the three previous months
21. Intensive exposure to sunlight or UV-rays on the studied zone within the previous month and/or foreseen during the study.
22. Subject planning to change her/his life habits during the study.
23. Subject with excessive consumption of alcohol (more than 2 glasses of wine per day) and/or tobacco (more than 10 cigarettes per day).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with cured wart after maximun 3 treatments evaluate by the investigator | Day 42

SECONDARY OUTCOMES:
Percentage of subjects with cured wart after 1, 2 and 3 treatments evaluated by the investigator common and plantar warts after 1, 2 and 3 treatments as assessed by the investigator | Day 14, Day 28, Day 42
Percentage of subjects with improved aspect of the wart after 1, 2 and 3 treatments evaluated by the investigator | Day 14, Day 28, Day 42
Mean frostbite area diameter after each treatment | Day 0, Day 14, Day 28
Percentage of subjects satisfied with the treatment by answering a questionnaire at the study end | Day 14, Day 28, Day 42
Illustration of the skin aspect by pictures before and after each treatment | Day 0, Day 14, Day 28
Mean subject' pain during treatment evaluated using a using a 11-item (0-10) Numerical Rating Scale | Day 0, Day 14, Day 28
  0= no pain; 10= worst possible pain
Subject tolerability evaluated at the study end by the investigator using a 4-item (0-3) Numerical scale | Day 14,Day 28, Day 42
  0=bad tolerance; 1= moderate tolerance; 2= good tolerance; 3 = very good tolerance
Collection of adverse events throughout the study | Day 0, Day 14, Day 28, Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Cegielska, MD, Principal Investigator — Dermascan
Locations (1):
- Eurofins Dermascan Poland, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No